CLINICAL TRIAL: NCT04740073
Title: Alterations in Muscle-tendon Mechanics and Contributions to Functional Change Prior to and Following Knee Replacement
Brief Title: How Muscle and Tendon Properties Contribute to Functional Change Prior to and Following Knee Replacement
Status: Suspended | Type: Observational
Why Stopped: Due to COVID-19 and research restrictions put in place by the university
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Jakobi, Principal Investigator, University of British Columbia
Other Study IDs: H18-02179
Record Dates: First submitted 2020-11-05; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Total Knee Arthroplasty
Keywords: Knee replacement; function; ultrasound; muscle; tendon; tendon mechanics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Persons undergoing total knee arthroplasty
- Controls: Persons not undergoing total knee arthroplasty who are age and sex-matched to the patient group.

SUMMARY:
It is unknown how progressive physiological change in muscle and tendon contributes to loss of functional ability in patients undergoing total knee replacement between referral to surgery, and during post-surgery recovery. This study will use ultrasound and neurophysiological measures to evaluate progressive alterations of tissue to understand functional decline in men and women prior to and following knee replacement surgery. A group of healthy controls not undergoing knee replacement will also be studied to contrast changes in the patient group to normal changes over time. It is hypothesized that from the point of referral to surgery, patients will exhibit reductions in muscle and tendon size (atrophy) and reflex excitability that will be greater in the surgical compared with non-surgical leg, and these changes will precede observable losses in functional measures and strength. Secondly, it is hypothesized that following total knee replacement, muscle and tendon size, reflex activity, strength and functional measures will increase to a level below the pre-surgery values.

DETAILED DESCRIPTION:
Osteoarthritis leads to degeneration of the articulating surfaces of the femur and tibia, with the end-stage intervention being replacement of these articulating surfaces using a total knee arthroplasty (TKA) surgical procedure. For patients undergoing TKA, there is a significant decline in functional abilities throughout the waiting period from surgical referral to the surgery date. Following the surgery, there is an improvement in function of these patients, but they do not reach the same functional level as healthy individuals who have not undergone TKA. To objectively measure functional abilities, various tests of strength, mobility and balance can be assessed. To date, no study has been conducted to evaluate how these objective measures of functional ability change throughout the pre-surgery waiting period and how this compares to levels following surgery. To gain a further understanding of the mechanisms behind these changes in function, physiological measures of muscle and tendon can be employed using electrical testing and ultrasound imaging. By evaluating changes in physiology alongside changes in function in TKA patients and healthy controls, we can gain a better understanding of the mechanisms underlying observable changes in function of patients undergoing TKA and how this compares to normal physiological changes in healthy controls.

Patients undergoing total knee replacement will visit the laboratory on 5 separate testing occasions (1, immediately following referral for TKA; 2, midpoint between referral and surgery; 3, 2 weeks prior to surgery; 4, 6 weeks post-surgery; 5, 6 months post-surgery. At each testing session participants will begin by filling out questionnaires related to overall functional ability. They will then perform functional tests of the upper and lower body to gain measures of limb-dependent functional ability. Following functional measures, resting measures of muscle and tendon surrounding the knee and quadriceps muscle group will be obtained using a combination of ultrasound imaging and measurements at the skin surface. Participants will then be equipped will surface electromyography (sEMG) electrodes on the muscles composing the quadriceps and hamstrings muscle groups to measure muscle activity during the subsequent measures. Muscle reflex activity will be assessed through sub-maximal and maximal electrical stimulation of the femoral nerve via carbon stimulation electrodes placed on the skin surface. Participants will then perform three maximal voluntary contractions (MVC) requiring them to extend their leg as hard as possible against the force transducer. Stimulation will be applied prior to, during and following the MVCs to assess the level of muscle activation. From the MVCs, sub-maximal tracking tasks of 5,10,25,50 and 75% MVC will be established. Using the force displayed on a screen in front of the participants, they will be required to produce contractions up to these force levels and maintain the force level for 5 second in order to quantify force steadiness. During these sub-maximal tracking tasks, the ultrasound probe will be placed on the junction between the quadriceps muscle and tendon to record tendon elongation for quantification of tendon mechanical properties.

These procedures will be preformed for the surgical leg of 30 patients undergoing TKA to compare inter-leg differences across time points, and 30 healthy control participants not undergoing TKA who are age-and sex-matched to the patient group will also perform these measures on their non-dominant leg using the same spacing between testing sessions. Measures will be compared between the surgical of patients and the non-dominant leg of healthy controls to evaluate differences over time in the patient group and how this compares to normal changes in a healthy population over the same period of time. This study will try and determine what measures of physiological change prior to surgery best predict optimization of patient function and improvement following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Referred by an orthopedic surgeon to undergo unilateral total knee arthroplasty,
* Age- and sex-matched controls who are not diagnosed with knee or hip osteoarthritis
* Read, speak and understand English

Exclusion Criteria:

* Prior replacement of a knee or hip joint
* Cardiometabolic or neurological disease beyond typical age-related decline
* Have had quadriceps tendon surgery
* Have had major and recent injury or surgery to either leg in prior 6 months
* Exclusion from electrical stimulation protocol if they have an implanted electronic device

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 patients undergoing unilateral total knee arthroplasty and 30 age- and sex-matched controls not undergoing total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in knee extension strength | Through study completion, an average of 1.5 years
  Maximal isometric knee extensions measured using a dynamometer by having participants push their shin against the dynamometer as hard as they can.

SECONDARY OUTCOMES:
Change in force steadiness | Through study completion, an average of 1.5 years
  Measure of one's ability to control force output of the knee extensors while tracing a target line displayed on the screen. Evaluated using the coefficient of variation of the force where a higher coefficient of variation is a less-steady contraction.
Change in Young's modulus | Through study completion, an average of 1.5 years
  Material property of the tendon consisting of tendon stiffness normalized to the tendon's dimensions (length and cross-sectional area). It is calculated as the slope of the stress-strain relationship where less tendon elongation with applied force leads to a higher Young's Modulus.
Change in timed up and go task | Through study completion, an average of 1.5 years
  Measure of one's ability to rise from a chair, walk a pre-defined distance to a cone, turn around the cone and return to the chair. Time is considered as the time from standing up form the chair until the participant is seated in the chair again. This measure provides an indication of dynamic balance control.
Change in balance | Through study completion, an average of 1.5 years
  Evaluating postural sway from a force platform during bipedal, tandem and single leg stance to determine participants' ability to balance across tasks with increasing difficulties. Participants will be required to maintain the stance as long as they can or until 60 seconds. Sway will be evaluated by analyzing the movement of the centre of pressure.

OTHER OUTCOMES:
Change in hand grip strength | Through study completion, an average of 1.5 years
  Handgrip strength measured by having participants squeeze a hand-held dynamometer. This provides an indication of overall strength.
Change in knee range of motion | Through study completion, an average of 1.5 years
  Used to evaluate mobility of the knee joint and participants' ability to voluntarily move the knee through its complete range of motion.
Change in 30-second chair rise | Through study completion, an average of 1.5 years
  The number of times a person can rise from a seated position in a chair to fully standing in 30-seconds. Provides a functional measure of muscle endurance.
Change in 36-item short form health survey (SF-36) score | Through study completion, an average of 1.5 years
  Questionnaire used to quantify health-status related to vitality, physical functioning, bodily pain, general health perceptions, physical, emotional, social roles and mental health. This questionnaire will be completed by both the patient group and the control group.
Change in Western Ontario and McMaster Universities osteoarthritis index (WOMAC) | Through study completion, an average of 1.5 years
  Questionnaire used to evaluate pain, disability and joint stiffness of the osteoarthritic joint. This questionnaire will only be completed by the patient group.
Change in Knee Injury and Osteoarthritis outcomes score (KOOS) | Through study completion, an average of 1.5 years
  Questionnaire used to assess the patient's opinion about their knee and associated problems. This questionnaire will only be completed by the patient group.
Change in muscle cross-sectional area | Through study completion, an average of 1.5 years
  Measurement of cross-sectional areas for the quadriceps and hamstrings muscle groups using ultrasound imaging. A static ultrasound image of the muscle in cross-section will be acquired and the border of the muscles will be traced to measure cross-sectional area. This measure provides an indication of changes in muscle size prior to and following surgery for the patient group. Muscle CSA will be measured for the control group to serve as a control comparison to the patient group.
Change in tendon length | Through study completion, an average of 1.5 years
  Measurement of lengths of the Quadriceps and Patellar tendons using ultrasound imaging. Images of the tendons will be obtained, and the length of the tendons will be measured from their muscle-tendon junction to the attachment of the tendon on the bone. Used to understand if there are changes in tendon length across the testing time frame or directly related to the surgery for the patient group, and the control group will serve as a control comparison.
Change in tendon cross-sectional area | Through study completion, an average of 1.5 years
  Measurement of tendon cross-sectional area for the quadriceps and patellar tendons using ultrasound imaging. A static ultrasound image of the tendon in cross-section will be acquired and the border of tendon will be traced to measured cross-sectional area. Used to understand if there are changes in tendon size across the testing time frame or directly related to the surgery for the patient group, and the control group will serve as a control comparison.
Change in muscle reflexes | Through study completion, an average of 1.5 years
  Muscle reflexes in the quadriceps evoked with electrical stimulation of the femoral nerve. Used to assess reflex feedback of the muscle with a larger reflex amplitude representing better reflex feedback.
Change in muscle activation | Through study completion, an average of 1.5 years
  Muscle activation will be assessed with surface electromyography for the quadriceps and hamstrings muscle groups to determine the amount of muscle activation required to execute the maximal and submaximal tracking tasks.
Change in tendon strain | Through study completion, an average of 1.5 years
  Tendon mechanical property quantified as elongation of the quadriceps tendon normalized to its resting length, and expressed as a percentage. This measure is obtained during the maximal and submaximal contractions using real-time ultrasound recordings of the muscle-tendon junction of the quadriceps and its tendon. The amount of elongation of the tendon during contraction is measured and this is normalized to the resting tendon length to obtain tendon strain.
Change in tendon stress | Through study completion, an average of 1.5 years
  Tendon mechanical property measured as the amount of force acting on the cross-sectional area of the tendon. This is calculated as the ratio of force to resting tendon cross-sectional area and provides an indication of the ability of the tendon to distribute load from the muscle.
Change in tendon stiffness | Through study completion, an average of 1.5 years
  Tendon mechanical property measured as the amount of tendon elongation for a given amount of applied force. This is calculated as the slope of the tendon force-elongation relationship, where a greater amount of force and lower amount of tendon elongation results in a steeper slope representing a stiffer tendon. Elongation is obtained using ultrasound imaging and force is the amount of force produced during the submaximal tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jakobi, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada